CLINICAL TRIAL: NCT03581331
Title: Consequence of Unilateral Vestibular Loss on Visual Abilities
Acronym: SVorthoptie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-45
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Vestibular Schwannoma; Visual Impairment; Vestibular Meniere Syndrome
MeSH Terms: conditions — Neuroma, Acoustic; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acute unilateral vestibular loss (Experimental): patients with acute unilateral vestibular loss by surgical deafferentation will performed an orthoptic balance
  Interventions: Diagnostic Test: orthoptic balance

INTERVENTIONS:
Diagnostic Test: orthoptic balance — Measurement of visual acuity by far: Monocular measurement, right eye, left eye and binocular Measurement of visual acuity closely: Monocular measurement, right eye, left eye and binocular Corneal reflection method or Hirschberg: Analysis of the corneal reflection after fixation of a point of fixation of light from a distance, then from near.
  Cover-Test: Study of the restitution movement following the fixation of the fixation point

SUMMARY:
Unilateral vestibular lesions are frequent and disabling pathologies causing a set of oculomotor, postural and perceptual symptoms. These symptoms reduce over time according to a vestibular compensation. However, vestibular compensation should be considered as a set of sub-processes whose duration and recovery level differ. Indeed, after a unilateral vestibular loss, some functions remain asymmetrical as a long-term effect, and these disorders may be observed among patients with no functional complaints. Balance disorders may persist in some patients.

The equilibration consists in handling real-time a considerable amount of information coming from the environment and the subject himself, allowing an adaptation of the position and movements of his body to satisfy the needs of posture, balance and orientation. This information comes mainly from the vision, the vestibule and the somesthesic system. It is pre-treated and harmonized in the brainstem, before being transmitted to the higher brain centres. Brain centers thus learn about peripheral conditions. According to these and the project of the movement, brain centers address in response orders to ophtalmological and motor effectors ensuring look, posture and balance to be provided. The eye is a cornerstone of the balancing system through the retina, an environmental sensor, and its extraocular muscles, effectors of the system.

The aim of this study is to assess the effects of acute unilateral vestibular loss on visual abilities evaluated by orthoptic balance in patients who presented acute unilateral vestibular loss by surgical deafferentation (removal of vestibular schwannoma, vestibular neurotomy or surgical labyrinthectomy for Meniere's disease), during the early phase and decline of vestibular compensation.

Our secondary objective is to evaluate the effect of a pre-existing anomaly of the visual abilities evaluated by orthoptic assessment on the vestibular compensation capacities.

All in all, this study seems crucial to improve the management of patients with unilateral vestibular dysfunction and contribute to improving their clinical management.

As a standardized management of these patients, an audio-vestibular evaluation will be performed before surgery (-1D), after acute unilateral vestibular loss at the early stage (+7D), and then after vestibular compensation (+2M) as well as an orthoptic evaluation. A good tolerance of the orthoptic evaluation is expected in this surgical context.

DETAILED DESCRIPTION:
Unilateral vestibular lesions are frequent and disabling pathologies, with significant psychological impacts, as well as on the socio-professional and daily life of the affected subjects. Furthermore, socio-economic consequences have to be considered.

The involvement of the vestibular system in the stabilization control of the look, the eye-head coordination, posture, locomotion and perception of verticality is widely recognized. Therefore, the unilateral vestibular diseases cause a set of oculomotor, postural and perceptual symptoms. These symptoms reduce over time according to a process known as vestibular compensation. However, vestibular compensation should be considered as a set of sub-processes whose duration and recovery level differ. Indeed, after a unilateral vestibular loss, some functions remain asymmetrical as a long-term effect, and these disorders may be observed among patients with no functional complaints. Balance disorders may persist in some patients.

The equilibration consists in handling real-time a considerable amount of information coming from the environment and the subject himself, allowing an adaptation of the position and movements of his body to satisfy the needs of posture, balance and orientation. This information comes mainly from the vision, the vestibule and the somesthesic system. It is pre-treated and harmonized in the brainstem, before being transmitted to the higher brain centres. Brain centres thus learn about peripheral conditions. According to these and the project of the movement, brain centers address in response orders to ophtalmological and motor effectors ensuring look, posture and balance to be provided. The eye is a cornerstone of the balancing system through the retina, an environmental sensor, and its extraocular muscles, effectors of the system.

The aim of this study is to assess the effects of acute unilateral vestibular loss on visual abilities evaluated by orthoptic balance in patients who presented acute unilateral vestibular loss by surgical deafferentation (removal of vestibular schwannoma, vestibular neurotomy or surgical labyrinthectomy for Meniere's disease), during the early phase and decline of vestibular compensation.

Our secondary objective is to evaluate the effect of a pre-existing anomaly of the visual abilities evaluated by orthoptic assessment on the vestibular compensation capacities.

All in all, this study seems crucial to improve the management of patients with unilateral vestibular dysfunction and contribute to improving their clinical management by prescribing an appropriate rehabilitation.

As a standardized management of these patients, an audio-vestibular evaluation (clinical ENT examination, pure tone and speech audiometry, videonystagmography, vestibular evoked myogenic potentials, Posturography, Vertical Visual Subjective, quality of life by Dizziness Handicap Inventory) will be performed before surgery (-1D), after acute unilateral vestibular loss at the early stage (+7D), and then after vestibular compensation (+2M).

An orthoptic evaluation will be performed during 30 min and the audio vestibular evaluation will be carried out at the same time. A good tolerance of the orthoptic evaluation is expected in this surgical context.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unilateral vestibular loss by programmed surgical deafferentiation: excision of vestibular schwannoma, vestibular neurotomy, or surgical labyrinthectomy for Meniere's disease
* Age between 18 and 80 years old.
* Women should not be pregnant or breastfeed; postmenopausal women can be included.
* A subject willing and able to give informed consent and to respect the requirements of the protocol.
* Affiliated with the French Social Security.

Exclusion Criteria:

* contralateral vestibular isflexia
* Central vestibular syndrome (stroke, intraparenchymal cerebral tumor, multiple sclerosis ...)
* Uni- or bilateral blindness
* Motor deficit
* Major medical or psychiatric illness that, in the opinion of the investigator, would pose a risk to or could compromise compliance with the study protocol.
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
orthoptic balance | 30 minutes
  orthoptic assessment

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France